CLINICAL TRIAL: NCT06890663
Title: The Use of Telehealth-Delivered Gut-Directed Hypnotherapy for Managing Gastrointestinal Health
Brief Title: Telehealth-Delivered Gut-Directed Hypnotherapy for Managing GI Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007687
Record Dates: First submitted 2025-03-20; First posted 2025-03-24 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Disease; Gastrointestinal Disorders; Nervous System
Keywords: Irritable Bowel Syndrome; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastrointestinal Diseases; Neurologic Manifestations; Irritable Bowel Syndrome; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Total enrollment time in the study will be 4 months. Participants will be divided into two groups of ten, and treatment will be provided in two 14-day intervention phases with one 3-month follow-up . One phase will include nonspecific hypnotherapy for relaxation, and one phase will include Gut-Directed Hypnotherapy (GDH) presented in a counterbalanced order depending on random assignment. Treatment conditions will be presented in a counterbalanced order depending on random assignment
  Hypnotherapy sessions will take place via Zoom sessions. There will be 4 sessions within each fourteen-day phase. Outcomes will be assessed through pre- and post-phase surveys, along with pre-and post-session surveys and one 3-month follow-up after completion of the two intervention phases.
  Interventions: Other: Nonspecific Hypnotherapy for Relaxation; Other: Gut-Directed Hypnotherapy (GDH); Other: 3-month Follow-Up
- Group 2 (Active Comparator): Total enrollment time in the study will be 4 months. Participants will be divided into two groups of ten, and treatment will be provided in two 14-day intervention phases with one 3-month follow-up . One phase will include nonspecific hypnotherapy for relaxation, and one phase will include Gut-Directed Hypnotherapy (GDH) presented in a counterbalanced order depending on random assignment. Treatment conditions will be presented in a counterbalanced order depending on random assignment
  Hypnotherapy sessions will take place via Zoom sessions. There will be 4 sessions within each fourteen-day phase. Outcomes will be assessed through pre- and post-phase surveys, along with pre-and post-session surveys and one 3-month follow-up after completion of the two intervention phases.
  Interventions: Other: Nonspecific Hypnotherapy for Relaxation; Other: Gut-Directed Hypnotherapy (GDH); Other: 3-month Follow-Up

INTERVENTIONS:
Other: Nonspecific Hypnotherapy for Relaxation — A therapeutic technique that uses hypnosis for relaxation.
Other: Gut-Directed Hypnotherapy (GDH) — A therapeutic technique that uses hypnosis and relaxation to help with gastrointestinal (GI) disorders.
Other: 3-month Follow-Up — A 3-month follow is completed after both intervention phases (general hypnotherapy and Gut Directed Hypnotherapy) are completed for each participant.

SUMMARY:
This study aims to evaluate the specific and non-specific effects of hypnotherapy and to evaluate the efficacy of group-format gut-directed hypnotherapy (GDH) delivered via telehealth for managing gastrointestinal health.

DETAILED DESCRIPTION:
Disorders of gut-brain interactions (DGBI) (also known as functional gastrointestinal disorders (FGID)) are defined as distinct combinations of chronic or recurrent gastrointestinal symptoms, with no obvious structural or biochemical abnormalities that explain symptomatology (Fairlieetal.,2023). DGBI symptoms are most likely generated based on a complex interaction among factors such as microbial dysbiosis within the gut, altered mucosal immune function, altered gut signaling (visceral hypersensitivity), and central nervous system dysregulation of the modulation of gut signaling and motor function (Drossman et al., 2016). Additionally, researchers have identified a bi-directional communication pathway between the central nervous system and the gastrointestinal (GI) tract, termed the gut-brain axis. The gut-brain axis suggests that changes in either the central nervous system or gut can disrupt the balance of the other. Therefore, psychosocial factors impacting the gut-brain axis increase GI symptoms and symptom severity and affect treatment outcomes (Vivier et al., 2020), and GI symptoms reduce psychosocial functioning in a reciprocal fashion.

The bi-directional communication system between the gut and brain is thought to play a critical role in maintaining gastrointestinal health and homeostasis, and an imbalance in either can have adverse consequences, often seen in conditions like IBS (Vivier et al., 2020). This is termed the gut-brain axis. It involves a complex interaction between the central nervous system (CNS) and the enteric nervous system (ENS), both of which regulate gut function and are affected by psychological states. Reflexes that generate appropriate gut responses to physiological as well as pathological afferent gut signals occur at the level of the ENS (Peters et al., 2015). Given this intricate connection, therapeutic approaches that target both physiological and psychological aspects may be particularly beneficial.

Based on the Rome IV criteria, there are several categories of DGBI including 1.) esophageal (e.g. gastroesophageal reflux disease (GERD, esophageal spasms)), 2.) gastroduodenal (e.g. chronic gastritis, peptic ulcer disease), 3.) bowel (e.g. irritable bowel syndrome (IBS), 4.) functional diarrhea), 5.) centrally mediated disorders of gastrointestinal (GI) pain (e.g. functional heartburn, functional abdominal pain syndrome (FAPS)), 6.) gallbladder and sphincter of oddie (e.g. sphincter of oddi dysfunction (SOD), biliary dyskinesia), 7.) anorectal (e.g. functional constipation, functional fecal incontinence), and 8.) childhood functional GI disorders (e.g. diarrhea, constipation, abdominal pain). A recent global internet survey of 54,127 adults across 26 countries found that 43% of people met the criteria for at least one FGID (Black et al., 2020). To date, there have not emerged highly effective interventions for these disorders, making it essential to explore innovative treatments. One such promising approach has been gut-directed hypnotherapy (GDH). The current study aims to evaluate (a) whether GDH offers symptom relief beyond the shared components of hypnotherapy and (b) the efficacy of GDH when delivered in group-based and telehealth formats. Findings will contribute to understanding GDH's role in DGBI management, in addition to its effectiveness in a group-based, telehealth format.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Self reported gastrointestinal symptoms consistent with disorders of gut-brain interaction
* English speaking
* Willingness to participate in all hypnotherapy sessions & complete all pre- and post-session surveys

Exclusion Criteria:

* Under 18 years
* Pregnant women
* Prisoners
* Children
* Individuals with active or a history of severe mental illness (e.g. active psychosis, dissociative disorders)
* A hypnotic susceptibility score in the low range (SHSS; total = 0-3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Patient- Reported Outcome Measurement Information System (PROMIS) | 4 months
  An NIH (National Institutes of Health)-funded initiative to develop and validate patient reported outcomes for clinical research and practice.
General Anxiety Disorder-7 (GAD-7) | 4 months
  A screening tool used to assess the severity of generalized anxiety disorder
Patient Health Questionnaire-9 (PHQ-9) | 4 months
  A self-administered questionnaire used to screen for and assess the severity of depressive symptoms
Patient Reported Outcome (PRO) | 4 months
  An assessment that directly captures a patient's self-reported health status, including their symptoms, quality of life, and functional ability, without interpretation from a healthcare provider

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cassisi, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States